CLINICAL TRIAL: NCT06663787
Title: Personalized Detection of ctDNA for Patients With HER2-Positive Metastatic Breast Cancer Who Achieved Durable Response by Anti-HER2 Treatment (HER2 CR)
Acronym: HER2 CR
Status: Active, not recruiting | Type: Observational
Sponsor: Nagoya City University (Other)
Responsible Party: Principal Investigator, Kazuki Nozawa, MD, Nagoya City University
Other Study IDs: HER2 CR; 80-24-0057 (Other: Nagoya City Unversity)
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer, Metastatic; HER2 + Breast Cancer
Keywords: ctDNA monitoring; MRD; minimal residual disease; HER2+ breast cancer; Dual response
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasm, Residual | interventions — Trastuzumab; Ado-Trastuzumab Emtansine; trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Continuing anti-HER2 treatment: Breast cancer patients who are continuing complete response (CR) or partial response (PR) for more than two years of anti-HER2 treatment (trastuzumab, pertuzumab, T-DM1, and T-DXd)
  Interventions: Drug: Trastuzumab (Herceptin); Diagnostic Test: SIgnatera
- Follow up (stop anti-HER2 treatment): Breast cancer patients who stopped anti-HER2 treatment with complete response (CR) or partial response (PR) after more than two years of anti-HER2 treatment(trastuzumab, pertuzumab, T-DM1, and T-DXd)
  Interventions: Diagnostic Test: SIgnatera

INTERVENTIONS:
Drug: Trastuzumab (Herceptin) — Continuing anti-HER2 treatment
  Other Names: Trastuzumab Emtansine; Trastuzumab Deruxtecan
  Groups: Continuing anti-HER2 treatment
Diagnostic Test: SIgnatera — A personalized, tumor-informed test.

SUMMARY:
Anti-HER2 therapy, such as trastuzumab and pertuzumab, has significantly improved long-term survival in HER2-positive breast cancer. The updated data of the CLEOPATRA trial showed significant Kaplan-Meier curves, suggesting the potential for a cure. However, the efficacy of maintenance therapy in long-term responders remains unexplored. This study will assess MRD in unresectable HER2-positive breast cancer cases with long-term response using the Signatera™ ctDNA assay, which could contribute to future treatment strategy development.

DETAILED DESCRIPTION:
More than 20 years have passed since the introduction of trastuzumab as a treatment for human epidermal growth factor receptor 2 (HER2)-positive breast cancer. The additive effect of trastuzumab, an anti-HER2 antibody, was evaluated in combination with chemotherapy (paclitaxel or anthracycline plus cyclophosphamide) in previously untreated, unresectable HER2-positive breast cancer. The number of cases achieving long-term survival with anti-HER2 therapy has been increasing, and this trend is also observed in our institution.

The treatment for unresectable breast cancer is systemic therapy, which is typically continued as long as it remains effective and side effects are tolerable. However, in cases of long-term response in HER2-positive breast cancer, the impact of continuing anti-HER2 therapy alone as maintenance therapy on prognosis and the safety of treatment discontinuation remains unclear.

In recent years, the clinical application of circulating tumor DNA (ctDNA) has attracted attention for early diagnosis and detection of minimal residual disease. Signatera™, an assay developed by Natera Inc., detects minimal residual disease. It is a personalized ctDNA test for individual patients, and a study targeting breast cancer patients post-surgery reported a detection sensitivity exceeding 90% for variant allele frequencies (VAF) as low as 0.01%. This high sensitivity has been reported not only in breast cancer but also in other cancer types. However, there have been no reports of Signatera analysis in unresectable breast cancer.

In this study, investigators will use Signatera™ to evaluate and analyze ctDNA status (ctDNA positive or negative) in cases of unresectable HER2-positive breast cancer that have achieved long-term response. By assessing ctDNA in such cases, this study may lead to new therapeutic strategies, such as de-escalating anti-HER2 therapy in ctDNA-negative cases.

ELIGIBILITY:
Inclusion Criteria:

* HER2 + metastatic breast cancer
* Pre / post menopausal
* Previously treated with anti-HER2 therapy
* Continuing CR or PR for more than 2 year

Exclusion Criteria:

* Patients who were deemed inappropriate as research subjects based on the physician's judgment, such as those possibly receiving inappropriate treatment.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligibility criteria for this study include patients who have been diagnosed with histologically confirmed invasive breast cancer and unresectable HER2-positive breast cancer. Eligible cases are those in which drug therapy, including anti-HER2 therapy, was initiated between January 1, 2000, and December 31, 2021. Additionally, patients must have maintained a partial or complete response to drug therapy, including anti-HER2 therapy, for more than two years. Finally, the study is limited to female patients aged 20 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The status of ctDNA | 1 year
  To assess the status of ctDNA in CR patients with/without continuing treatment, or PR patients with continuing treatment

CONTACTS AND LOCATIONS:
Locations (4):
- Natera, San Carlos, Texas, United States
- Japan (3):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Nagoya City University, Nagoya, Aichi-ken
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided